CLINICAL TRIAL: NCT03902873
Title: The Effect of a Real-time Audiovisual Feedback System on CPR Quality During In-hospital Cardiac Arrest: A Prospective Observational Study
Brief Title: The Effect of a Real-time Audiovisual Feedback System on CPR Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ho Geol Ryu, Associate professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: Audiovisual feedback_CPR
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Cardiopulmonary Resuscitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual compression (No Intervention): A group who get no real-time audiovisual feedback from the R Series® Monitor/Defibrillator (Zoll medical).
- real-time audiovisual feedback (Active Comparator): A group who get the real-time audiovisual feedback from the R Series® Monitor/Defibrillator (Zoll medical).
  Interventions: Other: Real-time audiovisual feedback

INTERVENTIONS:
Other: Real-time audiovisual feedback — During the chest compressions, doctors receive audiovisual feedback on the depth and speed of the appropriate chest compressions.
  Arms: real-time audiovisual feedback

SUMMARY:
The investigators will evaluate the effect of a real-time audiovisual feedback system on CPR quality during in-hospital cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 17 years old who require cardiopulmonary resuscitation in a medical or surgical intensive care units

Exclusion Criteria:

* Patients less than 18 years
* Patients with Do Not Resuscitate order
* Patients who require cardiopulmonary resuscitation outside a medical or surgical intensive care unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
chest compression fraction | 2 min
  the percentage of time in which chest compression are done by rescuers during a cardiopulmonary resuscitation

CONTACTS AND LOCATIONS:
Overall Officials: Ho Geol Ryu, Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Agree, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee H, Kim J, Joo S, Na SH, Lee S, Ko SB, Lee J, Oh SY, Ha EJ, Ryu HG. The effect of audiovisual feedback of monitor/defibrillators on percentage of appropriate compression depth and rate during cardiopulmonary resuscitation. BMC Anesthesiol. 2023 Oct 5;23(1):334. doi: 10.1186/s12871-023-02304-9. PMID 37798642